CLINICAL TRIAL: NCT00373126
Title: A Double-Blind, Placebo-Controlled Trial of Reward Responsivity During Nicotine Withdrawal in Smokers With Schizophrenia and Normal Controls
Brief Title: The Effects of Nicotine Withdrawal on Reward Responsivity in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: North Suffolk Mental Health Association (Other)
Collaborators: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CORRC 06-05; 2005P-001753
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: nicotine; schizophrenia; reward; withdrawal
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Tobacco Use Cessation Devices

INTERVENTIONS:
Drug: transdermal nicotine patch

SUMMARY:
It has been suggested that patients with schizophrenia smoke in order to produce amelioration of dysfunctional dopaminergic pathways allowing them to experience pleasure and satisfaction and overcome anhedonia. No studies have assessed the effects of nicotine withdrawal on reward responsivity in patients with schizophrenia. The investigators believe that an understanding of this is crucial if improved treatments for nicotine dependence are to be developed for this patient population. If this group already has deficits in reward responsivity as a symptom of the disease then they may be particularly prone to the effects of nicotine withdrawal on reward systems. Smoking cessation may lead to a further decrease in their responsivity to pleasurable stimuli and worsening anhedonia. Treatments for smoking cessation may need to ameliorate any increased deficits if they are likely to be effective in patients with schizophrenia.

DETAILED DESCRIPTION:
Heavy smoking continues to represent a significant public health problem for people in the general population and for people with major mental illness. Twenty-four percent of adults in the general population smoke and it has been estimated that 74-92% of people with schizophrenia smoke. While effective treatments for smoking cessation have been developed, response rates are modest and relapse rates are high. Approximately 70% of people who quit smoking with effective treatments relapse to smoking within one year. A syndrome of negative affect and anhedonia has been described as an important component in maintenance of dependence on nicotine. It has also been suggested that preventing the syndrome of anhedonia and negative affect during early abstinence may reduce relapse rates. If the syndrome of anhedonia can be measured objectively and quantitatively, we will be better able to test treatments for this withdrawal syndrome. It is our hypothesis that the syndrome of anhedonia during early abstinence from nicotine is quantifiable as a deficit in reward responsivity.

Animal studies suggest that nicotine withdrawal is associated with an alteration in reward responsivity. Brain stimulation reward thresholds have been used to measure anhedonia and responsivity to reward in animal models. Nicotine withdrawal has been associated with a significant decrease in brain reward function as measured by elevations in brain reward thresholds that persist for 4 days. Nicotine withdrawal has also been associated with failure of conditioning to an environment paired with novel stimuli, possibly due to a decrease in reward associated with novel stimuli. Drug withdrawal states have also been associated with inhibition of mesolimbic release in murine models.

We propose a randomized placebo controlled trial to investigate the effects of nicotine abstinence on reward responsivity in patients with no major mental illness and in patients with schizophrenia.

Principal Aims:

Aim 1: To evaluate the effects of nicotine withdrawal on a measure of reward responsivity Hypothesis 1a: Normal controls and subjects with schizophrenia will demonstrate deterioration on a measure of reward responsivity during abstinence (placebo condition) compared to baseline. (Primary Outcome Measure)

Aim 2: To evaluate the effects of transdermal nicotine on reward responsivity during abstinence.

Hypothesis 2a: Normal controls and subjects with schizophrenia will demonstrate greater response bias toward a rewarded condition following transdermal nicotine administration relative to placebo patch during a 3 day period of abstinence.

Aim 3: To evaluate the effects of smoking abstinence and transdermal nicotine on a measure of reward responsivity in patients with schizophrenia who smoke relative to normal control smokers.

Hypothesis 3a: Subjects with schizophrenia will demonstrate decreased reward responsivity during all conditions (baseline, nicotine replacement therapy condition and placebo condition) relative to normal controls.

Secondary aims:

Aim 4: To evaluate the effects of nicotine withdrawal on cognitive function in smokers Hypothesis 4a: Normal controls and subjects with schizophrenia will demonstrate poorer performance on tests of cognition following placebo administration compared with baseline and nicotine conditions.

We propose to test the effects of smoking abstinence and nicotine replacement therapy, using nicotine transdermal patch on a measure of reward responsivity in patients who smoke. We propose a randomized placebo controlled crossover trial with the primary outcome measure being Response bias using a signal detection task.

Subjects are 70 patients with schizophrenia who smoke and 70 normal control smokers who do not have a major mental illness and who are matched for age, sex and nicotine dependence. Though we expect to consent 70 subjects in each group, we expect only 20 subjects in each group to complete the study

ELIGIBILITY:
Inclusion Criteria:

Schizophrenia group inclusion criteria:

* DSM IV diagnosis of schizophrenia with stable symptoms and a stable dose of antipsychotic medications for at least 4 weeks
* Age 18-55 inclusive
* Able to provide informed consent
* Self reported smoking of 20 or more cigarettes per day for at least 12 months
* FTND score of >/= 5
* Expired air CO of >/= 10 ppm
* WRAT-3 IQ score greater than or equal to 35
* Normal or corrected to normal vision

Control group inclusion criteria: Same as above except for diagnosis of schizophrenia

Exclusion Criteria:

Schizophrenia Group exclusion criteria:

* Current unstable serious medical illness such as uncontrolled high blood pressure, untreated ischemic heart disease
* Use of any cholinesterase inhibitor such as galantamine in the past 3 months
* History of skin diseases (e.g., psoriasis), skin allergies, or strong reactions to topical preparations, medical dressings, tapes or nicotine patches
* Treated with an investigational medication in the last 30 days
* Currently or planning to become pregnant in the next 8 weeks as verified by positive pregnancy test or childbearing potential and not using adequate contraception
* Substance abuse in the past month: Self reported or diagnosed during chart review and verified by positive salivary test for cocaine, methamphetamine, amphetamine, ethanol, THC, opiates or PCP at screen
* Current major depressive disorder
* History of cognitive impairment due to other disorders such as head injury, dementia, general medical condition
* Diagnosis of mental retardation

Control group exclusion criteria: Same as above except for diagnosis of schizophrenia or family history of psychiatric illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-04

PRIMARY OUTCOMES:
Reward Responsivity using a signal detection task

SECONDARY OUTCOMES:
Cognitive drug research cognitive battery
Source monitoring task to assess verbal memory

CONTACTS AND LOCATIONS:
Overall Officials: A E Evins, MD MPH, Principal Investigator — North Suffolk Mental Health Association
Locations (1):
- Freedom Trail Clinic, 25 Staniford Street, Boston, Massachusetts, United States